CLINICAL TRIAL: NCT04885608
Title: Therapeutic Exercise for Older Adults: Revitalization and Postural Balance in Outdoor Fitness Parks
Brief Title: PReGe in Outdoor Fitness Parks
Acronym: PReGe-BIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Excelentísimo Ayuntamiento de Salamanca (Unknown)
Responsible Party: Principal Investigator, Fausto Jose Barbero-Iglesias, Dean, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PReGeUSAL-2021
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Frail Elderly
Keywords: Therapeutic exercise; Fraility; Functional capacity; Postural balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PReGe (Experimental): Group that will perform the intervention with therapeutic exercise.
  Interventions: Other: PReGe

INTERVENTIONS:
Other: PReGe — There will be two weekly sessions of 45 minutes, outdoors in outdoor fitness parks. The components of balance, gait, resistance, strength and elasticity will be worked on and breathing exercises will be performed. The sessions will be guided and dosed by physiotherapists, considering the level of perception of effort. Indications will be given to carry out other sessions of 60 to 120 minutes of therapeutic walking (minimum speed of 4 km/hour) during the week, to complete the 150-300 minutes per week of physical activity recommended by the WHO.

SUMMARY:
Older people have been one of the most affected by the Covid-19 pandemic. Restrictive measures to prevent the spread of the virus have affected the lifestyle of older people, which have reduced their level of physical activity. A sedentary lifestyle has negative health consequences, such as increased frailty and decreased functional capacity. The aim of the study is to apply a program of therapeutic exercise in outdoor fitness parks to prevent the complications of sedentary lifestyle. Community-dwelling older adults belonging will participate in an outdoor program to keep security measures and prevent contagion.

ELIGIBILITY:
Inclusion Criteria:

* People over 60 year who decide to participate voluntarily.
* Acceptance of Informed Consent.
* Municipal registration in Salamanca.
* Responsible declaration of good health.
* Absence of symptoms compatible with Covid-19.

Exclusion Criteria:

* Presence of absolute or relative contraindications to physical exercise.
* Presence of serious balance limitations, such as severe neurological, visual or musculoskeletal disorders.
* Presence of difficulties to carry out the tests of the Initial Assessment.
* Participate in another physical activity program.
* Incidents or pathologies suffered during the intervention that interfere with the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change from baseline to 16 weeks follow-up.
  A validated test to identify frail older adults. The score ranges from 0 to 12 points.
  The lowest scores are for people with the highest degree of frailty.
2 minute stair test | Change from baseline to 16 weeks follow-up.
  Test that evaluates cardiorespiratory endurance. There are reference tables that provide a percentile of resistance based on the age and gender of the participant.
Borg Rating of Perceived Exertion Scale | Change from baseline to 16 weeks follow-up.
  Exertion rating based on a 6 to 20 rating scale may provide a fairly good estimate of the actual heart rate during physical activity.
  Higher scores imply a greater degree of perceived exertion.
IPAQ-E Questionnaire | Change from baseline to 16 weeks follow-up.
  Questionnaire that evaluates the level of physical activity. The time spent on activities of different intensity during the last 7 days is recorded. The score is calculated in METs-minute-week (MMW). METs refer to a metabolic expenditure rate. A greater number of MMW, greater amount of physical activity is done weekly.

SECONDARY OUTCOMES:
Sex | Baseline
  Participant's sex will be registered.
Date of birth | Baseline
  Participant's date of birth will be recorded in order to calculate their age.
Medication | Baseline
  Information on the medication that each participant is currently taking will be collected to evaluate possible interferences.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto J Barbero-Iglesias, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided